CLINICAL TRIAL: NCT01705119
Title: The Effects of Vertical Position on Gas Exchange in Patients With Respiratory Failure
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12-1773
Record Dates: First submitted 2012-10-08; First posted 2012-10-12 (Estimated); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Respiratory Failure
Keywords: Mechanically Ventilated; Critical Care
MeSH Terms: conditions — Respiratory Insufficiency | interventions — Standing Position

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Mechanically Ventilated (Experimental)
  Interventions: Other: Standing

INTERVENTIONS:
Other: Standing

SUMMARY:
The purpose of this study is to investigate how changing from a supine to upright position affects gas exchange for patients with hypoxemic respiratory failure.

The research question is: will oxygen saturation and/or partial pressure of oxygen in the blood change when a patient with hypoxemic respiratory failure moves from a supine to upright position?

DETAILED DESCRIPTION:
Our hypothesis is that blood oxygen tension will not decrease and may even increase when a patient with respiratory failure stands up. Supine positioning often causes partial lung collapse, which results in a decreased amount of lung being available for gas exchange. In patients with Acute Respiratory Distress Syndrome (ARDS), tilting the patient up in bed has been shown to increase oxygen tension and improve lung compliance. Positional changes are sometimes used as a "rescue" intervention in patients with severe hypoxemia from ARDS. The investigators hope to conclude that severe hypoxemia should not be viewed as a contraindication to physical therapy, but rather physical therapy may be a potential intervention for patients with marginal gas exchange.

After sedative interruption, physical therapists and nursing staff will assist mechanically ventilated patients in moving to the side of the bed. They will assess the extremity strength using the MRC scale. If lower extremity strength is at least 4/5, the patient will be assisted to assume the upright position. The investigators will monitor the patient continuously and the session will be stopped at any point for

A. Mean arterial pressure <65 B. Heart rate <40, >130 beats/min C. Respiratory rate <5, >40 breaths/ min D. Pulse oximetry <88% E. Marked ventilator dyssynchrony F. Patient distress G. New arrhythmia H. Concern for myocardial ischemia I. Concern for airway device integrity J. Endotracheal tube removal

At this point, the patient's vital signs, pulse oximetry, and measures of lung compliance will be obtained. If an arterial line is in place and there have been ventilator adjustments since the morning arterial blood gas, the investigators will draw an arterial blood gas.

The physical therapists and nursing staff will then help the patient stand up. After one minute, the investigators will record another set of vital signs, pulse oximetry, and measures of lung compliance from the mechanical ventilator. If an arterial line is in place, the investigators will draw another arterial blood gas.

The patient will then be assisted back into bed. One hour later, the investigators will record the patient's vital signs, pulse oximetry, and measures of lung compliance from the mechanical ventilator.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ≥18 years who are mechanically ventilated
* An oxygen saturation of 88-94% or an arterial line

Exclusion Criteria:

* Mean arterial pressure <65
* Heart rate < 40 or > 130 beats/min
* Respiratory rate < 5 or > 40 breaths/min
* Pulse oximetry < 88%
* Evidence of elevated intracranial pressure
* Active gastrointestinal blood loss
* Active myocardial ischemia
* Pregnancy
* Actively undergoing a procedure
* Patient agitation requiring increased sedative administration in the last 30 mins
* Insecure airway (device)
* The patient was not ambulatory prior to hospitalization
* The patient's body habitus and/or mental status make it unsafe to stand up
* The patient has been placed on strict bed rest by the treating physicians

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2012-10-01 (Actual); Primary Completion 2021-06-10 (Actual); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
PaO2 to FiO2 ratio | change from baseline to 1 hr

SECONDARY OUTCOMES:
Oxygen Saturation | change from baseline to 1 hr
change in blood PCO2 | change from baseline to 1 hr
Change in blood pH | change from baseline to 1hr

OTHER OUTCOMES:
Tidal Volume | change from baseline to 1 hr
Vital Signs | change from baseline to 1hr

CONTACTS AND LOCATIONS:
Overall Officials: John P Kress, MD, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago Medical Center, Chicago, Illinois, United States